CLINICAL TRIAL: NCT02269345
Title: Auricular Acupuncture: A Novel Application in Ureteral Stent Pain.
Brief Title: Auricular Acupuncture in Ureteral Stent Pain
Acronym: AAstent
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unworkable. This study had several PIs and attempted several avenues of recruitment. Still were only able to recruit 34 out of the 120 needed.
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FWH20140088H
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Battlefield Acupuncture (Experimental): BFA at points cingulate gyrus, thalamus, omega 2, shen-men, point zero
  Interventions: Other: Battlefield Acupuncture
- Standard Treatment (Placebo Comparator): Standard Treatment alone
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Other: Battlefield Acupuncture — Battlefield Acupuncture at points cingulate gyrus, thalamus, omega 2, shen-men, point zero
  Arms: Battlefield Acupuncture
Other: Standard Treatment — Standard Treatment alone.
  Arms: Standard Treatment

SUMMARY:
The investigators propose to complete a randomized controlled trial to compare battlefield auricular acupuncture at five points in right ear and five points in left ear (cingulate gyrus, thalamus, omega 2, point zero, and shen men) plus standard of care, versus standard of care alone, for symptomatic treatment of stent pain in postoperative ureteral stent patients. Male and female DoD beneficiaries ages 18 years or older, who are scheduled for elective urologic surgery that would be expected to have the routine placement of a ureteral stent (ureteroscopy, ureteroscopy with biopsy, ureteroscopy with laser treatment of a stone, ESWL of stone greater than 10mm) will be recruited. Subjects will be followed up at 24 hours post surgery, 48 hours, 1 week, 1 month, and 1 month post surgery. The investigators will ask subjects to rate their pain level on a 0-10 analogue scale, the investigators will assess via the Ureteric Stent Symptoms Questionnaire (USSQ) subjects' urinary urgency, urinary frequency, and quality of life. The investigators will ask subjects how many pills they have taken for their pain including the quantity and dose to assess a reduction in pain medication use.

DETAILED DESCRIPTION:
Subjects will be ages 18 years or older and scheduled for routine urologic surgery. To randomize subjects, the investigators will employ a random number generator, which will minimize difference between study groups.

Screening Visit:

Obtain signed Informed Consent document and HIPAA Authorization. Review past medical history in Armed Forces Health Longitudinal Technology Application (AHLTA) to verify the inclusion/exclusion criteria including previous encounter, vital signs review, medication list, co-morbidities, prior surgical history, demographics, problems list, and note any prior acupuncture received.

Subjects will be given a Medication Log to assist them in documenting the amount of pain medications that they are taking as part of standard of care.

Subjects will be given a handout of standard BFA Discharge Instructions including what an infection looks like and what to do in the event of an infection (see attached).

Visit 1 (Baseline):

Subjects will be randomized into 1 of 2 groups:

Group 1: Standard operative and standard post-operative care plus BFA (up to 5 acupuncture needles* in each ear at points cingulate gyrus, thalamus, omega 2, shen-men, point zero, identified by point-finder) Group 2: Standard treatment alone. Subjects will be given treatment according to their randomization group. The investigators review the subject's medical record and document any standard of care pain assessments that were performed upon admission and after pain intervention to the Post Anesthesia Care Unit (PACU) and Same Day Surgery Unit (SDSU). The investigators will also record the amounts of standard of care pain medications used during their hospital stay.

All subjects, regardless of randomization group, will be instructed to have no heavy meals, no excessive hot or cold foods, no heavy exercise or intercourse, and no alcohol for 24 hours after Visit 1.

Ear Acupuncture needles will fall out on their own within about one week.

Visit #2 (24 hours post-surgery):

Subject will be contacted in-person, via phone, email, or text message asked:

On a scale of 0-10, with 10 being the worst pain, what is their pain level? Have they returned to work or resumed normal household duties? If so, how many hours post-surgery? What pain medication are they taking? And what strength? How many total doses have they taken since their surgery? Essentris electronic inpatient medical record will be reviewed to determine total dose of pain medications received if still in hospital.

Is the patient voiding without irritative symptoms? Urinary frequency, urgency, dysuria, hematuria will be assessed.

Visit #3 (48 hours post- surgery)

Subject will be contacted either in-person, or via phone, email or text message and asked:

On a scale of 0-10, with 10 being the worst pain, what is their level of pain? Have they returned to work or resumed normal household duties? If so, how many hours post-surgery? What pain medication are they taking? And what strength? How many total doses have they taken since their surgery? Essentris electronic inpatient medical record will be reviewed to determine total dose of pain medications received if still in hospital.

Is the patient voiding without irritative symptoms? Urinary frequency, urgency, dysuria, hematuria will be assessed.

Visit #4 (1 week post-surgery)

Subject will be contacted either in-person, or via phone, email or text message and asked:

Have they returned to work or resumed normal household duties? If so, how many days post-surgery? What pain medication are they taking? And what strength? How many total doses have they taken since their surgery? USSQ (Stent in Situ) will be administered to patients.

Visit #5 Visit (1 month post surgery with stent in-situ or 5 weeks post stent removal at week 1)

Subject will be contacted either in-person, or via phone, email or text message and asked:

Have they returned to work or resumed normal household duties? If so, how many days post-surgery? What pain medication are they taking? And what strength? How many total doses have they taken since their surgery? USSQ (Post Stent) will be administered to patients.

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion:

* Male and female DoD beneficiaries
* Age 18 years or older who are scheduled for elective urologic surgery that would be expected to have the routine placement of a ureteral stent (ureteroscopy, ureteroscopy with biopsy, ureteroscopy with laser treatment of a stone, extracorporeal stone wave lithotripsy (ESWL) of stone greater than 10mm).

Exclusion:

* Pregnant or breastfeeding.
* Traumatic ureteral injury repairs with stents.
* Ureteral stents placed during procedures for urologic cancer treatments.
* Sepsis prior to stent placement or other active urologic infection.
* Absence of ear.
* Active cellulitis of ear.
* Ear anatomy precluding identification of acupuncture landmarks.
* Non-English speaking.
* Use of Hearing Aids that preclude the insertion of ASP needles.
* Inability to comply with study protocol.
* Patients receiving treatment for chronic pain conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
improved ability to tolerate the presence of the ureteral stent | 1 month
  This will be assessed via the Ureteric Stent Symptoms Questionnaire

SECONDARY OUTCOMES:
reduce narcotic use | 1 month
  We will ask the participant during each visit what pain medication are they taking? And what strength? How many total doses have they taken since their surgery?
post-operative readmission rates for pain/irritative symptoms | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, MD, Principal Investigator — Mike O'Callaghan Federal Medical Center
Locations (1):
- Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No